CLINICAL TRIAL: NCT05434923
Title: PORTHOS - PORTuguese Heart Failure Observational Study: a Nationwide Epidemiological Study on Heart Failure and Asymptomatic Left Ventricle Systolic Dysfunction Based on Contemporary Diagnostic Tools
Brief Title: PORTHOS - PORTuguese Heart Failure Observational Study
Acronym: PORTHOS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Sociedade Portuguesa de Cardiologia (Unknown); NOVA Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: D1699R00015
Record Dates: First submitted 2022-06-08; First posted 2022-06-28 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
Keywords: Prevalence; Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the prevalence of heart failure in the resident population in mainland Portugal aged 50 years or above, using a contemporary, guideline-based diagnostic approach, to optimize patient management and improve strategic healthcare decision-making

DETAILED DESCRIPTION:
The contemporary prevalence of heart failure in Portugal is largely unknown and may differ from that reported in early studies, which were conducted in the late 1990s-early 2000s with the diagnostic techniques available at the time and did not include neither advanced echocardiographic parameters nor natriuretic peptides measurements. Thus, a large and representative study is needed to address knowledge gaps on the epidemiology, characteristics and burden of heart failure in Portugal. The study aims to determine the prevalence of global heart failure, as well as heart failure subtypes. It also aims to assess the distribution of comorbidities among patients with heart failure, as well as patients' health-related quality of life. The Investigators will conduct a population-based study with a three-stage design approach, enrolling 5616 subjects aged 50 years or above, randomly selected through multi-stage sampling, using the National Health Service as reference: PHASE 0 - Participant selection/enrollment through phone call; PHASE 1 - Screening (NT-proBNP levels determination), health-related quality of life evaluation and sociodemographic characterization; PHASE 2 - Confirmatory assessment with a 12-lead electrocardiography, comprehensive transthoracic echocardiography, extended symptoms assessment and biomarkers assessment; PHASE 3 - Heart failure with preserved ejection fraction exertion testing through a non-invasive echocardiographic diastolic stress test.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling citizens living in Mainland Portugal;
* Registration in a primary care centre;
* Age ≥50 years at recruitment;
* Voluntary signed informed consent.

Exclusion criteria:

* Living in institutions (e.g., nursing homes, prisons, military facilities, hospitals);
* Non-Portuguese speakers;
* Reduced physical and/or cognitive ability hampering participation (e.g., blindness, deafness, or cognitive impairment).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community dwelling adults aged 50 years and above living in Mainland Portugal and registered in the National Health Service patients' database. Population will be stratified by age and gender.
Sampling Method: Probability Sample
Enrollment: 6189 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of HF among the mainland resident Portuguese population aged 50 or above. | Between March 2022 and March 2023
  Prevalence of HF among the mainland resident Portuguese population aged 50 or above.

SECONDARY OUTCOMES:
Age- and gender-specific prevalence of HF among the Portuguese population. | Between March 2022 and March 2023
  Age- and gender-specific prevalence of HF among the Portuguese population.
Heart Failure reduced Ejection Fraction phenotype prevalence. | Between March 2022 and March 2023
  Heart Failure reduced Ejection Fraction phenotype prevalence.
Heart Failure mildly reduced Ejection Fraction phenotype prevalence | Between March 2022 and March 2023
  Heart Failure mildly reduced Ejection Fraction phenotype prevalence
Heart Failure preserved Ejection Fraction phenotype prevalence. | Between March 2022 and March 2023
  Heart Failure preserved Ejection Fraction phenotypes prevalence.
Prevalence of asymptomatic NT-proBNP elevation. | Between March 2022 and March 2023
  Prevalence of asymptomatic NT-proBNP elevation.
Prevalence of Pre-HF, as defined by the HF universal definition 2, in patients with asymptomatic NT-proBNP elevation. | Between March 2022 and March 2023
  Prevalence of Pre-HF, as defined by the HF universal definition 2, in patients with asymptomatic NT-proBNP elevation.
Prevalence of comorbidities among Portuguese HF patients | Between March 2022 and March 2023
  Prevalence of comorbidities among Portuguese HF patients, namely:
  1. CHD,
  2. previous MI,
  3. hypertension,
  4. obesity,
  5. DM,
  6. VHD,
  7. AF,
  8. CKD,
  9. COPD,
  10. OSA;
Prevalence of comorbidities among patients with HFrEF, HFmrEF, and HFpEF phenotypes. | Between March 2022 and March 2023
  Prevalence of comorbidities among patients with HFrEF, HFmrEF, and HFpEF phenotypes, namely:
  1. CHD,
  2. previous MI,
  3. hypertension,
  4. obesity,
  5. DM,
  6. VHD,
  7. AF,
  8. CKD,
  9. COPD,
  10. OSA.
Health-related quality of life 5-level Euro Quality of life-5D version (EQ-5D-5L) | Between March 2022 and March 2023
  Health-related quality of life 5-level Euro Quality of life-5D version (EQ-5D-5L) consists of 2 pages: the descriptive system (EQ-5D) and the visual analogue scale (EQ VAS).
  EQ-5D comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression; each one has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0).
Health-related quality of life (Kansas City Cardiomyopathy Questionnaire - KCCQ) | Between March 2022 and March 2023
  Health-related quality of life (Kansas City Cardiomyopathy Questionnaire - KCCQ).
  The predictor was the annually updated KCCQ score. The KCCQ is a validated instrument to assess health status among persons with heart failure. The self-administered questionnaire includes 23-items which quantify the importance of dyspnea, fatigue, and edema on physical, social, and emotional functions. The responses are categorized under 3 subscales (symptom burden, physical limitation and quality of life) with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The total KCCQ score represents the mean of the three subscale scores.
Association between health-related quality of life questionnaire (EQ-5D-5L) results and the HF phenotype. | Between March 2022 and March 2023
  Association between health-related quality of life questionnaire (EQ-5D-5L) results and the HF phenotype.
Association between health-related quality of life questionnaire (KCCQ) results and the HF phenotype. | Between March 2022 and March 2023
  Association between health-related quality of life questionnaire (KCCQ) results and the HF phenotype.

OTHER OUTCOMES:
Exploratory Outcome: Association between pre-diabetes and HF prevalence. | Between March 2022 and March 2023
  Association between pre-diabetes and HF prevalence.
Exploratory Outcome: Association between diabetes mellitus and HF prevalence. | Between March 2022 and March 2023
  Association between diabetes mellitus and HF prevalence.
Exploratory Outcome: Association between biomarkers of interest (HbA1c%) and HF prevalence. | Between March 2022 and March 2023
  Association between biomarkers of interest (HbA1c%) and HF prevalence.
Exploratory Outcome: Association between biomarkers of interest (serum creatinine) and HF prevalence. | Between March 2022 and March 2023
  Association between biomarkers of interest (serum creatinine) and HF prevalence.
Exploratory Outcome: Association between biomarkers of interest (C-reactive protein) and HF prevalence. | Between March 2022 and March 2023
  Association between biomarkers of interest (C-reactive protein) and HF prevalence.
Exploratory Outcome: Association between biomarkers of interest (troponin) and HF prevalence. | Between March 2022 and March 2023
  Association between biomarkers of interest (troponin) and HF prevalence.
Exploratory Outcome: Association between biomarkers of interest (lipids) and HF prevalence. | Between March 2022 and March 2023
  Association between biomarkers of interest (lipids) and HF prevalence.
Exploratory Outcome: Association between biomarkers of interest (HF biomarkers) and HF prevalence. | Between March 2022 and March 2023
  Association between biomarkers of interest (HF biomarkers) and HF prevalence.
Exploratory Outcome: Distribution of HF according to geographical area using NUTS II segmentation. | Between March 2022 and March 2023
  Distribution of HF according to geographical area using NUTS II segmentation.

CONTACTS AND LOCATIONS:
Locations (13):
- Portugal (13):
  - Research Site, Aljustrel
  - Research Site, Aveiro
  - Research Site, Braga
  - Research Site, Castelo Branco
  - Research Site, Coimbra
  - Research Site, Lagos
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Serpa
  - Research Site, Setúbal
  - Research Site, Silves
  - Research Site, Sobral de Monte Agraço
  - Research Site, Torres Vedras

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1699R00015&attachmentIdentifier=da13d09b-3a7b-4622-b2fd-a259a18bff66&fileName=redacted_CSR.pdf&versionIdentifier=